CLINICAL TRIAL: NCT02707211
Title: Immunization Against oxLDL in Patients With Lysosomal Lipid Diseases and Associated Metabolic Disorders
Brief Title: Anti-oxLDL IgM Antibodies as a Novel Therapy for Metabolic Lipid Diseases
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Annick Vanclooster, Nurse, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pfizer-Prevenar13-2015
Record Dates: First submitted 2016-01-20; First posted 2016-03-14 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Lipid Metabolism, Inborn Errors
MeSH Terms: conditions — Lipid Metabolism, Inborn Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-oxLDL IgM antibodies (Experimental): administration Anti-oxLDL IgM antibodies
  Interventions: Biological: Anti-oxLDL IgM antibody

INTERVENTIONS:
Biological: Anti-oxLDL IgM antibody — Immunization

SUMMARY:
To test whether active pneumococci immunization can alleviate inflammation and improve cholesterol metabolism in lysosomal lipid storage diseases and associated metabolic disorders.

DETAILED DESCRIPTION:
Growing evidence describes the central role of oxidized low density lipoproteins (oxLDL) in diseases related to lipid metabolism. Moreover, oxLDL has been shown to be involved in pathological processes such as an inappropriate inflammatory response, disturbance of cholesterol metabolism and dysfunction of the lysosomal apparatus. Relevantly, it has been shown that immunizing mice with Streptococcus pneumoniae results in higher serum titers of anti-oxLDL IgM antibodies due to molecular mimicry.

ELIGIBILITY:
Inclusion Criteria:

* Patients of following diseases (characterized by lysosomal lipid storage or associated metabolic pathology)

  * Familial hypercholesterolemia,
  * NPB,
  * NPC
  * Partial lipodystrophy (PPARg mutations and laminin A/C mutations)
* Intention to be treated and participate to the treatment - Written informed consent

Exclusion Criteria:

* Medical conditions that may interfere with the study procedures: cancer Hodgkin lymphoma (all related to immune cells); autoimmune diseases; immune deficiency; splenectomy syndrome
* Alcohol abuse (quantitative limit >20g/day for men and >10g for women)
* Illiteracy
* Patients younger than 10 years.
* Any condition which in the opinion of the (co-) investigator might interfere with the evaluation of the study objectives.

Ages: 2 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
The level of inflammation | 4 weeks

SECONDARY OUTCOMES:
Levels of lysosomal enzymes | 4 weeks
the level of cholesterol metabolism | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided